## **Official Title:**

Factors Associated with the Quality of Life of Nursing Home Residents in Vietnam: A Cross-Sectional Study

**NCT Number:** Pending

**Date of Document:** September 2025

#### **INFORMED CONSENT FORM**

# Factors Associated with the Quality of Life of Nursing Home Residents in Vietnam: A Cross-Sectional Study

| MonthDate Year |
|---|
| 1. Study Participants Older adults aged 60 years and above who are currently residing in nursing homes in Hanoi and some neighboring provinces in Northern Vietnam, who are able to communicate and understand the questionnaire, and who agree to participate in the study. Study Location: |
| 2. Confirmation of Having Read and Understood the Study Information Sheet We invite you to participate in this study by answering a questionnaire through a face-to-face interview. Please carefully read the Study Information Sheet provided together with this Conser Form. Please check (X) the appropriate box: ☐ I have read and clearly understood the contents of the Study Information Sheet/Protocol ☐ I have not read |
| 3. Confirmation of Voluntary Participation I confirm that I voluntarily agree to participate in this study, and I understand that I may refusor withdraw from the study at any time without affecting my rights at the nursing home. I understand that during the study, if the survey results show that I may have abnormal signs related to physical or mental health (e.g., severe depression, serious memory impairment), the research team may refer me to medical staff or related specialists at the facility where I reside/work, for further monitoring and support. This referral is only intended to ensure my health and safety, is not mandatory, and I have the full right to refuse if I do not wish to receive such support. |
| 4. Confirmation of Audio Recording (if applicable) ☐ I agree to allow audio recording during the interview for research purposes, with the assurance of confidentiality. ☐ I do not agree to audio recording. |
| 5. Confirmation of Participation in the Study Please check (X) the appropriate box: ☐ I agree to participate in the study ☐ I do not agree to participate in the study |

### **6.** Contact Information of the Principal Investigator

Name: Nguyễn Thị Thu Trang

Address: School of Nursing, National Taipei University of Nursing and Health Sciences

Email: trangseri@gmail.com Phone: +84 354 858 599

### 7. Contact Information of the Ethics Committee (for questions/complaints)

Ethics Committee - Hanoi University of Public Health

Address: No. 1A, Duc Thang Road, Dong Ngac Ward, Hanoi, Vietnam

Phone: +84 24 6266 3024 Email: <u>irb@huph.edu.vn</u>

CONFIRMATION OF PARTICIPANT (Signature and Full Name)

CONFIRMATION OF RESEARCHER (Signature and Full Name)

Nguyễn Thị Thu Trang